CLINICAL TRIAL: NCT03434327
Title: The Comparative Impacts of Power Training and Strength Training Programs on Neuromuscular Performance and Other Physical Measurements in Individuals With Parkinson's Disease
Brief Title: Training and Parkinson's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180001
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Parkinson Disease; Weight-Lifting Exercise Program
MeSH Terms: conditions — Parkinson Disease | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training (Experimental): Strength training will use 75-80% of the subject's maximum for the specific exercise and contractions will occur at 2s concentric and 3s eccentric. All training will be performed on Keiser air-driven machines. Subjects will perform 10 exercises targeting all major muscle groups. The training will last for12 consecutive weeks, for a total of 24 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes warm-up, 50 minutes of training and five minutes of cool-down.
  Interventions: Other: Strength Training
- Power Training (Experimental): For power training the subjects will perform the concentric phase at high speed, while eccentric portion will last approximately 2 sec. Loads will vary from 30-80% of the subject's maximum depending on the biomechanical nature of the joints involved in the exercise. All training will be performed on Keiser air-driven machines. Subjects will perform 10 exercises targeting all major muscle groups. The training will last for 12 consecutive weeks, for a total of 24 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes warm-up, 50 minutes of training and five minutes of cool-down.
  Interventions: Other: Power Training

INTERVENTIONS:
Other: Strength Training — Eleven resistance training exercises performed on pneumatic resistance training machines using 2 second concentric and 3 second eccentric contractions at 75-80% of each subjects maximal strength. Subjects will perform 3 sets per exercise, two times per week for 12 weeks.
  Arms: Strength Training
Other: Power Training — Eleven resistance training exercises performed on pneumatic resistance training machines using maximum speed concentric and 3 second eccentric contractions at the load that produces the highest power for the individual. Subjects will perform 3 sets per exercise, two times per week for 12 weeks.
  Arms: Power Training

SUMMARY:
The purpose of the current study is to compare the impacts of specifically designed power training and strength training programs on function and physical performance in Parkinson's patients. Specific aims are to examine the impact of these interventions on performance variables such as balance, strength, power, posture, gait and physical function.

DETAILED DESCRIPTION:
This study will look at how well two different training programs (strength and power training) do at improving the participant's physical functions. Before and after training, the participant will go to our laboratory on four separate days for screening and testing.

Approximate time schedules for each day are provided below:

Day 1 0:00-0:40: Informed consent meeting Mini-mental test, and Health Status Questionnaire, Hoehn & Yahr Classification of Disability for PD, UPDRS motor examination and PQ-39.

Details regarding study participation will be explained and the participant will be provided the opportunity to ask questions about the study as well as being informed that the participant have the right to end participation at any time without consequence. In addition, this time will be used to identify if the participant can safely take part in the study.

0:40-0:41: Randomization of intervention The participant will successively pull one piece of paper out of a bowl. Each piece of paper will have one of the two intervention programs on it.

0:41-0:46: Anthropometric Measurements The participant's height and weight will be measured using a standard mechanical physician's scale with a height rod. In addition, the participant's blood pressure will be measured using our automated system.

0:46-0:70: Familiarization with the tests Details of each field test including the Berg Balance Test, TUG, the standard proprioception test on the Proprio 5000, muscle power and strength, the Dynamic Gait Analysis (DGI), and 3D gait and tremor analysis be explained to the participant. The participant will be allowed to practice the tests under our guidance and will be allowed to ask any questions at this time.

Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination

The participant's speech, facial expression, tremor, rigidity, posture, gait, and slowness of body movement will be observed and rated by a trained researcher during the course of other assessment activities and certain other items will be specifically tested by that researcher. These activities include:

* rapid hand movement,
* gait initiation and gait,
* rising from chair and
* response to sudden posterior pull on shoulders while standing. .

Day 2 0:00-0:05: The Falls Efficacy Scale (FES) This will be used to determine the participant's level of self-efficacy (how the participant feels about himself or herself) as it relates to fear of falling.

The FES takes about 5 minutes to complete and consists of questions related to the participant's concern about the possibility of falling when the participant do 10 specific daily living activities (ADL).

0:05-0:20: The Berg Balance Scale.

The Berg Balance Scale is a 14-item test designed to measure the participant's standing balance while the participant are standing still and moving. The test takes about 15-20 minutes and tests the following activities:

Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers, Standing with eyes closed, Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, and Standing on one foot.

0:20-0:25: Recovery period

0:25-0:35: The Timed Up and Go Test (TUG) The participant will be asked to stand up from a standard chair with a seat height of between 40 and 50 cm, walk a 3-m distance at a normal pace, turn, walk back to the chair, and sit down. The test takes approximately 2-4 minutes to complete with instructions.

0:35-0:40: Recovery period

0:40-0:55: The Dynamic Posturography Test (Proprio 5000) The participant will complete a dynamic balance test on a moving platform that rocks around at different speeds and angles and tests how well the participant can keep the participant's balance. For the participant's safety the participant will wear a harness that is attached to the machine so that the participant cannot fall.

Day 3 0:00-0:30: Muscle strength and Power Examination.

Measurements will be taken during:

* Chest Press (pushing the machine handles away from the chest like the participant do in a push-up),
* Seated Rows (pulling the machine handles toward the body, like rowing a boat)
* Lat Pulldowns (bringing the machine handles down toward the participant's shoulder)
* Shoulder Press (pushing the machine handles upward away from the participant's shoulder)
* Biceps curl (bring the handles up by bending the elbows, like "making a muscle")
* Triceps pushdown (pushing the handles straight down starting with the elbows bent and handles at the waist)
* Leg Press (sitting with legs bent and pushing outward)
* Calf Raises (toe pushdown),
* Hip adduction (pushing both legs inward toward the center line of the participant's body)
* Hip abduction (pushing both legs outward away from the center line of the participant's body) Muscle strength and power will be assessed using air resistance rather than plates. To determine strength, one-repetition maximum (1RM) will be measured for each muscle group. The participant will perform the concentric phase within the limits of the participant's own specific range of motion for each joint/movement tested over 2 s periods. The tester will gradually increase the resistance for each repetition until the participant are not able to move the lever arm one time through the full ROM. The participant will be asked how hard the test felt after each repetition and each muscle group will be finished in a maximum of seven repetitions.

0:30-0:40: Recovery Period

0:50-0:90: Power test After measurement of the participant's strength for each movement, we will measure the participant's power using the same machines. The participant's power will be assessed at 40%, 50%, 60%, 70%, 80%, or 90% of the participant's maximum strength depending on the exercise. Before performing each exercise, the participant will be instructed to perform the exercises as fast as possible through the full ROM. A 3-minute rest will be provided between exercises. Three trials will be performed per exercise and the highest power recorded will be designated as the participant's peak power.

Day 4 0:00-0:20: Gait Test: The gait test will be a standard 10m gait test at usual (two trials) and maximum (2 trials) speed. The participant will be timed using a wireless infrared timing system and movement analysis will be performed using our 3D movement analysis system and force plates.

0:20-0:25: Recovery Period 0:25-0:40: Hand tremor will be tested using an infrared camera. The participant will then be asked to turn over five coins and button the front of a shirt. These tests will be timed.

Training program After the pre-testing of the study is done, the participant will come to the lab twice a week for 12 consecutive weeks, for a total of 24 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes warm-up, 50 minutes of the training program to which the participant have been randomly assigned and five minutes of cool-down. The training programs will be a power training program and a standard strength program.

All training will be performed on our Keiser air-driven machines. Subjects will perform 10 exercises including:

Chest Press Seated Rows Lat Pulldowns Shoulder Press Biceps curl Triceps pushdown Leg Press Calf Raises Hip adduction Hip abduction And perform 3 sets of 12-15 repetitions of each exercise,

Both programs will begin with low resistance/speed training with gradual increases for the first two weeks and then progress to the specific program.

Strength training will use 75-80% of the subjects maximum for the specific exercise and contractions will occur at 2s concentric and 3s eccentric. For power training the subjects will perform the concentric phase at high speed, while eccentric portion lasts approximately 2 sec.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 89 years old, Hoehn & Yahr Classification of Disability, stage 1-3 who can ambulate with or without an assistive device for at least 50 feet and are able to get up and down from the floor with minimal assist or less. A score of 24 or above on the Folstein Mini-Mental State Exam.

Exclusion Criteria:

* Stage greater than 4 on the Hoehn & Yahr Classification of Disability, decline in immune function such as pneumonia or systemic infection, progressive degenerative disease besides PD, spinal fusion or other orthopedic surgery in the past six months, mental disease/psychosis such as dementia, greater than minimal assistance required for gait and transfers, inability to make regular time commitments to the scheduled training sessions, or in a resistance training program within the past year

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG) | 2-4 minutes
  The participant will be asked to stand up from a standard chair with a seat height of between 40 and 50 cm, walk a 3-m distance at a normal pace, turn, walk back to the chair, and sit down. The test takes approximately 2-4 minutes to complete with instructions.
Strength Test | 30 minutes
  The participant will perform the concentric phase within the limits of the participant's own specific range of motion for each joint/movement tested over 2 s periods. The tester will gradually increase the resistance for each repetition until the participant are not able to move the lever arm one time through the full ROM. The participant will be asked how hard the test felt after each repetition and each muscle group will be finished in a maximum of seven repetitions.
Power test | 30 minutes
  After measurement of the participant's strength for each movement, we will measure the participant's power using the same machines. The participant's power will be assessed at 40%, 50%, 60%, 70%, 80%, or 90% of the participant's maximum strength depending on the exercise. Before performing each exercise, the participant will be instructed to perform the exercises as fast as possible through the full ROM. A 3-minute rest will be provided between exercises. Three trials will be performed per exercise and the highest power recorded will be designated as the participant's peak power.
Gait Test | 20 minutes
  The gait test will be a standard 10m gait test at usual (two trials) and maximum (2 trials) speed. The participant will be timed using a wireless infrared timing system and movement analysis will be performed using our 3D movement analysis system and force plates.

SECONDARY OUTCOMES:
The Falls Efficacy Scale (FES) | 5 minutes
  This will be used to determine the participant's level of self-efficacy (how the participant feels about himself or herself) as it relates to fear of falling.
Berg Balance Scale. | 15-20 minutes
  The Berg Balance Scale is a 14-item test designed to measure the participant's standing balance while the participant are standing still and moving. The test takes about 15-20 minutes and tests the following activities:
  Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers, Standing with eyes closed, Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, and Standing on one foot.
Dynamic Posturography Test | 5 minutes
  The participant will complete a dynamic balance test on a moving platform that rocks around at different speeds and angles and tests how well the participant can keep the participant's balance. For the participant's safety the participant will wear a harness that is attached to the machine so that the participant cannot fall.
Manual dexterity | 15 minutes
  Hand tremor will be tested using an infrared camera. The participant will then be asked to turn over five coins and button the front of a shirt.

CONTACTS AND LOCATIONS:
Locations (1):
- Max Orovitz Laboratories, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No